CLINICAL TRIAL: NCT03731533
Title: WellStart Type 2 Diabetes Study
Brief Title: WellStart Reboot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grantor withdrew from study
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-X-292
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; lifestyle; nutrition; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention group will be enrolled in WellStart. The control group will continue with usual care. Study subjects from both groups will be sent commercial home lab kits to test lipid and hemoglobin A1c levels, as well as a digitally connected scale and blood pressure monitoring device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WellStart (Experimental): WellStart is a 12-week virtual intensive therapeutic lifestyle program utilizing web-based encounters with physicians, dietitians, health coaches and additional resources.
  Interventions: Behavioral: WellStart
- Usual Care (No Intervention): The control group will continue with usual care.

INTERVENTIONS:
Behavioral: WellStart — 1. Five weekly automated text messages linked to an online article on health and wellness.
  2. Five weekly automated health coach motivational text message to smart phone. Optional back and forth text with their health coach is available.
  3. Daily Option to participate and post comments or questions in online discussion forum moderated by health coaches.
  4. Three group (up to 20 participants) health coach online visits (60 minutes).
  5. Two online group visits with a dietitian in groups of 10-12 participants.
  6. Three one-on-one online visits with a Physician Advisor to review progress, review any changes in medications by the primary medical provider (PCP), review biometrics and lab results, review safety guidelines and symptoms (30 minutes).
  Arms: WellStart

SUMMARY:
This is a randomized, controlled comparison study that will evaluate the effectiveness of WellStart, a virtual intensive therapeutic lifestyle change program to control type 2 diabetes.

DETAILED DESCRIPTION:
Purpose: To test the efficacy of WellStart Health program to to arrest and / or reverse type 2 diabetes.

Future comparative studies between programs programs are anticipated, utilizing this data to help identify the strengths and weaknesses of different programs, as well as identify subpopulations that might benefit from one program as opposed to another.

Data from this study will be shared via posters and papers among the lifestyle medicine community / publications to help contribute to better lifestyle interventions.

Pilot programs reported on the WellStart web page report reduction in hemoglobin A1c (HBA1c) and weight during the 12 week program.

The web site states:

Evidence for the Program:

The 12-week lifestyle medicine program provides online health coaching and education on 5 domains of wellbeing: whole food, plant-forward nutrition, movement, mindset and social support and resilience. The pilot programs have shown a mean weight reduction of 6.9 lbs in 85% of participants of the 12-week program. 85% of participants with prediabetes experienced a reduction in hemoglobin A1c, while 100% of those with diabetes had a mean hemoglobin A1c reduction of 1.1. WellStart has also helped 35% of participants on pharmacotherapy, eliminate medication (antihypertensives and metformin).

Studies have shown the ability of plant-based nutrition to reverse chronic disease including coronary artery disease. The BROAD study found a statistically significant reduction in BMI and cholesterol in those following a plant-based diet. Furthermore, Dean Ornish's research showed regression of coronary atherosclerosis after 5 years of a plant-based diet in addition to lifestyle changes and found that it reduced cardiac events by half. Caldwell Esselstyn's research on a whole food plant-based diet also demonstrated a significant reduction in major cardiac events in adherent patients.

Furthermore, a 2016 comprehensive literature review supports a plant-based diet as medical nutrition therapy for diabetes based on its ability to reduce fasting blood glucose, hemoglobin A1c, body mass index and reduce medication use.

The Diabetes Prevention Program (DPP), a lifestyle and diet intervention program, reduces the risk of diabetes by half in a population at risk. It has been successfully adapted to the online setting. WellStart is taking this concept a step further by providing participants with additional education and support to transition to plant-forward nutrition habits.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type 2 diabetes (T2DM)
* Between the ages of 18 and 65 years-old
* Own and willing to use a smart phone or computer, and have daily internet access
* Have an email account
* Have access to resources (finances and transportation) that allow for regular acquisition (at least once weekly) of groceries, including produce
* Access to resources that allow for food preparation at home (refrigeration, basic kitchen appliances and supplies)
* Willingness to attempt changes in food preparation and consumption, and physical activity.

-Scoring at least a 7/10 in both readiness for change and confidence of success; 1= not ready / no confidence; 10 = extremely ready / extremely confident of success -

Exclusion Criteria:

* Dementia
* Advanced renal disease (stage 4 or 5) with or without hemodialysis
* Congestive Heart Failure
* Taking warfarin
* Pregnancy or plans for pregnancy
* Current smoker of tobacco cigarettes
* Adults who have a physical limitation to prepare their own food or incorporate movement into their lifestyle (based on questionnaire answer)
* Brittle diabetes and/or history of hospitalization for high or low blood sugar
* Difficult-to-control hypertension and / or on 4 or more medications for high blood pressure.
* Does not speak or understand English
* Inability to use email or the Internet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months
  glycosylated hemoglobin, measure of diabetes control over last 3 months
Weight | 6 months
  risk factor for diabetes

SECONDARY OUTCOMES:
Short Form Health Survey - 36 Questions (SF-36) | 6 months
  Survey of patient health status
Total cholesterol | 6 months
  risk factor for cardiovascular disease, a comorbidity of diabetes
Low density lipoprotein cholesterol (calculated) | 6 months
  risk factor for cardiovascular disease, a comorbidity of diabetes
High density lipoprotein cholesterol | 6 months
  risk factor for cardiovascular disease, a comorbidity of diabetes
Triglycerides | 6 months
  risk factor for cardiovascular disease, a comorbidity of diabetes
Systolic Blood Pressure | 6 months
  risk factor for cardiovascular disease, a comorbidity of diabetes
Diastolic Blood Pressure | 6 months
  risk factor for cardiovascular disease, a comorbidity of diabetes
Days per week of exercise | 6 months
  Average days per week of exercise, self reported by patient
Minutes per day of exercise | 6 months
  Average minutes per day of exercise, self reported by patient

CONTACTS AND LOCATIONS:
Overall Officials: David S Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song M, Fung TT, Hu FB, Willett WC, Longo VD, Chan AT, Giovannucci EL. Association of Animal and Plant Protein Intake With All-Cause and Cause-Specific Mortality. JAMA Intern Med. 2016 Oct 1;176(10):1453-1463. doi: 10.1001/jamainternmed.2016.4182. PMID 27479196
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] Esselstyn CB Jr. Updating a 12-year experience with arrest and reversal therapy for coronary heart disease (an overdue requiem for palliative cardiology). Am J Cardiol. 1999 Aug 1;84(3):339-41, A8. doi: 10.1016/s0002-9149(99)00290-8. PMID 10496449
- [Background] Diabetes Prevention Program Research Group; Knowler WC, Fowler SE, Hamman RF, Christophi CA, Hoffman HJ, Brenneman AT, Brown-Friday JO, Goldberg R, Venditti E, Nathan DM. 10-year follow-up of diabetes incidence and weight loss in the Diabetes Prevention Program Outcomes Study. Lancet. 2009 Nov 14;374(9702):1677-86. doi: 10.1016/S0140-6736(09)61457-4. Epub 2009 Oct 29. PMID 19878986